CLINICAL TRIAL: NCT06442878
Title: Effects of Psychomotor Intervention Program Mediated by Belly Dance in Adults Women.
Brief Title: Benefits of a Belly Dance Psychomotor Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Simone Leara Barroso Pereira, MS, University of Évora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UÉ
Record Dates: First submitted 2024-05-30; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Adult Women
Keywords: woman, body awareness, dance, balance and well-being.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control and Experimental Group (Other): The same group, will do the intervention will attend the belly dance program. The control group will maintain the usually daily activities, not attending any exercise program for a month and a half, and than will be a experimental group with 2 sessions / week of 60 minutes on alternated days.
  Interventions: Other: Belly Dance Program

INTERVENTIONS:
Other: Belly Dance Program — All Belly Dance sessions comprised 5 phases: 1) opening ritual (5 min), in which participants will be welcomed and perceived how people were feeling. 2) warm-up (15 min), in which thinking and feeling are integrated during the movements, isolating each part of the body according to Laban's body organization. 3) main phase (30 min), will be proposed individual, pair and group activities, in order to achieve the objectives planned. This phase will end with a choreography composition or a challenge; 4) cool-down (5 min) with stretching and physiological parameters normalization; and 5) ending ritual (5 min), in which the participants will be invented to share their sessions' experience.

SUMMARY:
The aim of the present study is to analyze the effects of a psychomotor intervention program mediated by belly dance in adult women. This Quasi-experimental study is a controlled trial with one arm. Participants will be allocated to one group which will be i) control and ii) experimental. That is at first i) will attend a control period without intervention (6 weeks) and at second ii) will attend an intervention period participating on the intervention program mediated by belly dance (12 weeks). Participants will be accessed at a baseline, at post control and at post intervention.

DETAILED DESCRIPTION:
Sedentary lifestyles has been identified as one of the main causes for the development of pathologies as are cardiovascular diseases and of mental health problems such as anxiety and depression. Associated with this, psychomotor factors can also be negatively affected as well as the perception of well-being. Women's daily life associated with tasks accumulation is referred to as a barrier to engaging in physical have progressively made it more difficult for them to perform formal physical activity (Barranco-Ruiz, 2020). Dance can help in this scenario because it is a pleasurable activity that favors social and intrapersonal relationships, working simultaneously on factors such as balance, motor coordination, agility, body awareness, and rhythm, having a positive impact on quality of life and well-being. In this way, dance, through its various components associated with movement, can assume a character of health promotion, also making possible a space of attention for women (Hernandes et al, 2018). Studies have already been carried out focusing on the effects of belly dancing on body image, quality of life and self-esteem in women with cancer, experienced and professional experienced and professional belly dancers/practitioners, elderly women with depression, pregnant women and depression, pregnant women and those with chronic pain (Boing, 2018; Toberna, 2020; Castrillon, 2017). No studies were found that looked at psychomotor factors (balance, agility and body body awareness), or indicators of well-being focused on body image, movement image and and mood states.

The proposed study has a quasi-experimental design with two pre-tests and one post- test, with only one group, the experimental group being its own control. In this way, we will apply Pre-test 1 and after six weeks without intervention, we will apply Pre-test 2 in order to obtain the results referring to the control group. After that, we will start the intervention itself, which will last twelve weeks and will culminate with the Post test 1.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged > 17 years and <60 years
* Availability to participate in the program

Exclusion Criteria:

* Presence of cognitive impairment (Mini-Mental State Examination);
* Presence of motor impairment, neurological problems or diseases compromising the program participation;
* Unavailability to participate in the program.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to post control and to post intervention | [ 0, 6 weeks] vs. [0,12 weeks]
  Balance and Postural Control outcome measure assessed by Modified Star Excursion Balance Test (MSEBT); stand stork test and standing stork test (blind).
Change from Baseline to post control and to post intervention | [ 0, 6 weeks] vs. [0,12 weeks]
  Agility outcome measure assessed by Hexagonal Obstacle Test.
Change from Baseline to post control and to post intervention | [ 0, 6 weeks] vs. [0,12 weeks]
  Rhythm perception and reproduction assessed by Go No Go Test
Change from Baseline to post control and to post intervention | [ 0, 6 weeks] vs. [0,12 weeks]
  Body Awareness outcome measure assessed by the Multidimensional Assessment of Interoceptive Awareness (MAIA), ranging an 8-scale state-trait questionnaire with 32 items and the Awareness-Body-Chart test (ABC).
Change from Baseline to post control and to post intervention | [ 0, 6 weeks] vs. [0,12 weeks]
  Body Image outcome measure will assessed using the Body Investment Scale (BIS), ranging with a Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Change from Baseline to post control and to post intervention | [ 0, 6 weeks] vs. [0,12 weeks]
  Image of movement outcome measure will accessed using the miq-3 test, made up of three subscales to assess the kinesthetic and visual modalities; and two Likert-type subscales with 7 levels of response, ranging from "very difficult" to "very easy".
Change from Baseline to post control and to post intervention | [ 0, 6 weeks] vs. [0,12 weeks]
  Mood States outcome measure will accessed using the Poms Mood Test with a likert scale with a score of 0 "not at all" and 5 "very much".

CONTACTS AND LOCATIONS:
Locations (1):
- Simone Leara Barroso Pereira, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barranco-Ruiz Y, Paz-Viteri S, Villa-Gonzalez E. Dance Fitness Classes Improve the Health-Related Quality of Life in Sedentary Women. Int J Environ Res Public Health. 2020 May 26;17(11):3771. doi: 10.3390/ijerph17113771. PMID 32466496
- [Result] Boing L, Baptista F, Pereira GS, Sperandio FF, Moratelli J, Cardoso AA, Borgatto AF, de Azevedo Guimaraes AC. Benefits of belly dance on quality of life, fatigue, and depressive symptoms in women with breast cancer - A pilot study of a non-randomised clinical trial. J Bodyw Mov Ther. 2018 Apr;22(2):460-466. doi: 10.1016/j.jbmt.2017.10.003. Epub 2017 Oct 12. PMID 29861250
- [Result] Castrillon T, Hanney WJ, Rothschild CE, Kolber MJ, Liu X, Masaracchio M. The effects of a standardized belly dance program on perceived pain, disability, and function in women with chronic low back pain. J Back Musculoskelet Rehabil. 2017;30(3):477-496. doi: 10.3233/BMR-150504. PMID 27858690
- [Result] Hernandes JC, Di Castro VC, Mendonca ME, Porto CC. Quality of life of women who practice dance: a systematic review protocol. Syst Rev. 2018 Jul 10;7(1):92. doi: 10.1186/s13643-018-0750-5. PMID 29991355
- [Result] Toberna CP, Horter D, Heslin K, Forgie MM, Malloy E, Kram JJF. Dancing During Labor: Social Media Trend or Future Practice? J Patient Cent Res Rev. 2020 Apr 27;7(2):213-217. doi: 10.17294/2330-0698.1723. eCollection 2020 Spring. PMID 32377554